CLINICAL TRIAL: NCT01477450
Title: Comparison of Oxygen Delivery Devices for Reversal of Altitude-Induced Hypoxemia in Normal Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rich Branson, M.D., Clinical Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Branson-2010-02
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Hypoxemia; Hypobaric Hypoxemia
Keywords: Hypobaric hypoxemia; Altitude; Oxygen; oxygen concentrator
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 L/min ; 16 mL (Active Comparator): Cylinder oxygen delivery (1 L/min) followed by pulse-dose oxygen by concentrator (16 mL)
  Interventions: Device: Pulse-dose oxygen; Device: Cylinder oxygen delivery
- 2 L/min ; 32 mL (Active Comparator): Cylinder oxygen delivery (2 L/min) followed by pulse-dose oxygen by concentrator (32 mL)
  Interventions: Device: Pulse-dose oxygen; Device: Cylinder oxygen delivery
- 3 L/min ; 48 mL (Active Comparator): Cylinder oxygen delivery (3 L/min) followed by pulse-dose oxygen by concentrator (48 mL)
  Interventions: Device: Pulse-dose oxygen; Device: Cylinder oxygen delivery

INTERVENTIONS:
Device: Pulse-dose oxygen — Pulsed-dose oxygen delivery from an oxygen concentrator
Device: Cylinder oxygen delivery — Oxygen delivery from an oxygen cylinder

SUMMARY:
This study will compare the ability of pulsed-dose oxygen from a concentrator to reverse altitude-induced hypoxemia compared to compressed gas from a standard oxygen cylinder.

DETAILED DESCRIPTION:
Subjects will be monitored non-invasively with pulse oximetry, end-tidal carbon dioxide, tissue oxygenation and ECG. The mean seal level oxygen saturation will be recorded.Subjects exposed to an altitude of 14,000 feet will experience moderate hypobaric hypoxia. The mean oxygen saturation at this altitude is 83%. Subjects will receive oxygen from both an oxygen concentrator or a cylinder of oxygen following exposure to hypobarism. Oxygen from each source will be increased in 1 liter per minute increments until the oxygen saturation returns to the baseline sea level oxygen saturation.

The oxygen requirement to return oxygen saturation to baseline values will be recorded. The flow from the concentrator and the cylinder will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Current altitude chamber certification
* Age 18 years - 60 years

Exclusion Criteria:

* Current upper respiratory infection
* Current symptoms of lower respiratory infection -- productive cough

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Branson, MSc RRT, Principal Investigator — University of Cincinnati
Locations (1):
- Brooks City Base, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 L/Min ; 16 mL | 2 L/Min ; 32 mL | 3 L/Min ; 48 mL
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 L/Min ; 16 mL | 2 L/Min ; 32 mL | 3 L/Min ; 48 mL | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Customized [Number; unit: participants]
  18-65 years | 10 | 10 | 10 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 6
  Male | 9 | 7 | 8 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 6 | 11
  Not Hispanic or Latino | 6 | 9 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Return of Oxygen Saturation to Baseline (Sea Level) Values
Description: Oxygen will be titrated from either an oxygen concentrator or an oxygen cylinder in liters per minute until the oxygen saturation returns to the sea level value. The flow in liters per minute is the dependent variables. Each participant will experience induced hypoxemia followed by cylinder oxygen delivery; each will also experience induced hypoxemia followed by pulse-dose oxygen from a concentrator.
Time Frame: 50 minutes
Measure: Number; unit: participants
Arm/Group | 1 L/Min ; 16 mL | 2 L/Min ; 32 mL | 3 L/Min ; 48 mL
Number analyzed (Participants) | 10 | 10 | 10
participants
  Reversal of hypoxemia after pulse-dose oxygen | 6 | 8 | 10
  Non-reversal of hypoxemia after pulse-dose oxygen | 4 | 2 | 0
  Reversal of hypoxemia after cylinder O2 delivery | 9 | 10 | 10
  Non-reversal of hypoxemia after cylinder O2 delive | 1 | 0 | 0
Statistical Analysis 1: Comparison: 1 L/Min ; 16 mL; Test type: Superiority or Other; p = 0.3, Chi-squared
Statistical Analysis 2: Comparison: 2 L/Min ; 32 mL; Test type: Superiority or Other; p = 0.47, Chi-squared
Statistical Analysis 3: Comparison: 3 L/Min ; 48 mL; Test type: Superiority or Other; p = 1.00, Chi-squared

ADVERSE EVENTS:
Arm/Group | 1 L/Min ; 16 mL | 2 L/Min ; 32 mL | 3 L/Min ; 48 mL
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes